CLINICAL TRIAL: NCT05552573
Title: A Randomized, Blinded, Positive-controlled Phase I Clinical Trial to Evaluate the Safety and Immunogenicity of Recombinant SARS-CoV-2 Vaccine (CHO Cell) LYB001 in Population Aged 18 Years and Above
Brief Title: Safety and Immunogenicity of COVID-19 Vaccine in Population Aged 18 Years and Above
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Guangzhou Patronus Biotech Co., Ltd. (Industry)
Collaborators: Yantai Patronus Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LYB001/CT-CHN-101
Record Dates: First submitted 2022-09-15; First posted 2022-09-23 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2022-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low-dose vaccine(18-59 years) (Experimental): 3 doses of LYB001 or Recombinant COVID-19 Vaccine (CHO Cell) at the immunization schedule of 0, 28, 56 days. Vaccination or positve-controlled group will be randomly assigned to receive in a 4:1 ratio.
  Interventions: Biological: low-dose LYB001; Biological: Recombinant COVID-19 Vaccine (CHO Cell)
- Low-dose vaccine(60 years old and above) (Experimental): 3 doses of LYB001 or Recombinant COVID-19 Vaccine (CHO Cell) at the immunization schedule of 0, 28, 56 days. Vaccination or positve-controlled group will be randomly assigned to receive in a 4:1 ratio.
  Interventions: Biological: low-dose LYB001; Biological: Recombinant COVID-19 Vaccine (CHO Cell)
- High-dose vaccine(18-59 years) (Experimental): 3 doses of LYB001 or Recombinant COVID-19 Vaccine (CHO Cell) at the immunization schedule of 0, 28, 56 days. Vaccination or positve-controlled group will be randomly assigned to receive in a 4:1 ratio.
  Interventions: Biological: Recombinant COVID-19 Vaccine (CHO Cell); Biological: high-dose LYB001
- High-dose vaccine(60 years old and above) (Experimental): 3 doses of LYB001 or Recombinant COVID-19 Vaccine (CHO Cell) at the immunization schedule of 0, 28, 56 days. Vaccination or positve-controlled group will be randomly assigned to receive in a 4:1 ratio.
  Interventions: Biological: Recombinant COVID-19 Vaccine (CHO Cell); Biological: high-dose LYB001

INTERVENTIONS:
Biological: low-dose LYB001 — This vaccine is prepared through gene recombination and 3 doses of low-dose(30µg/0.5ml) LYB001 at the schedule of 0, 28, 56 days.
  Arms: Low-dose vaccine(18-59 years); Low-dose vaccine(60 years old and above)
Biological: Recombinant COVID-19 Vaccine (CHO Cell) — This vaccine is Positive-controlled vaccine and 3 doses (0.5ml) at the schedule of 0, 28, 56 days.
Biological: high-dose LYB001 — This vaccine is prepared through gene recombination and 3 doses of high-dose(60µg/0.5ml) LYB001 at the schedule of 0, 28, 56 days.
  Arms: High-dose vaccine(18-59 years); High-dose vaccine(60 years old and above)

SUMMARY:
This is a randomized, blinded, positive-controlled study to evaluate the safety and immnunogenicity of Recombinant SARS-CoV-2 Vaccine (CHO Cell) LYB001, in population aged 18 years old and above. 100 subjects will be recruited in this study, including 50 aged 18-59 years old and 50 aged 60 years old and above.

DETAILED DESCRIPTION:
All subjects will be received 3 doses of LYB001, according to the immunization schedule of 0, 28, 56 days. The adverse events within 28 days after vaccination will be observed. In addition, blood samples will be collected on day 0 before vaccination,day 14 after dose 2, and on day 14, 28 and month 3, 6, 9, 12 after full vaccination. Serum antibody levels, cellular immune responses will be analyzed to evaluate the immunogenicity and immune persistence of the vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and above.
* Participate the trial voluntarily and sign informed consent form.
* Subjects are willing to comply with the requirements of the clinical trial protocol -and complete the study follow-up.
* Armpit temperature ≤37.0℃ on the day of enrollment.
* Novel Coronavirus (COVID-19) Antibody (IgG and IgM) was negative.

Exclusion Criteria:

* Known allergy to investigational vaccine or its excipients, or previous history of anaphylactic shock or other serious adverse reactions to other vaccines
* History of severe acute respiratory syndrome (SARS) and/or Middle East respiratory syndrome (MERS) infection or disease;
* History of COVID-19, or close contact with a confirmed/suspected COVID-19 patient, or SARS-CoV-2 nucleic acid test was positive or antibody test (IgG, IgM) was positive;
* Used antipyretic drugs, painkillers or anti-allergic drugs within 24 h before enrollment;
* Has received COVID-19 vaccine;
* vaccination of subunit vaccines and/or inactivated vaccines within 7 days before enrollment, or vaccination of live attenuated vaccines within 14 days before enrollment;
* Administration of blood or blood related products (including immunoglobulins) within 3 months before enrollment; or plan to use during the trial;
* Patients with the following diseases:

  1. Any acute disease or in the acute phase of chronic diseases within 7 days before enrollment;
  2. Congenital malformation or developmental disorder, genetic defect, severe malnutrition, etc.;
  3. History of congenital or acquired immunodeficiency or autoimmune diseases, or long-term(used continuously>14 days)use of glucocorticoid (dose ≥ 20 mg/day prednisone or equivalent dose) or other immunosuppressants within the last 6 months, yet the following situations are allowed to be included: inhaled or topical use of external steroids, or short-term use (course ≤ 14 days ) of oral corticosteroids;
  4. Known diagnosis of or having infectious diseases, or positive for any one of HBsAg, anti-HCV antibody, anti-TP antibody or anti-HCV antibody;
  5. Neurological diseases or family history (convulsion, epilepsy, encephalopathy, etc.); history of psychosis or family history;
  6. Asplenia or functional asplenia;
  7. Serious or uncontrollable cardiovascular diseases, diabetes, hematological and lymphatic diseases, immune system diseases, liver and kidney diseases, respiratory diseases, metabolism and bone diseases, or malignant tumors that need hospitalization;
  8. Contraindications of intramuscular injection and blood drawing, such as coagulation dysfunction, thrombosis or hemorrhagic diseases, or any condition that needs continuous use of anticoagulant;
  9. Severe hypertension with uncontrolled medication (at field measurement: systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥100mmHg) History of major surgery within 12 weeks before enrollment (in the opinion of the investigator), or incomplete recovery after surgery, or planning major surgery during the trial;
* Participating or will participate other clinical trials during this trial;
* Any disease or condition that, in the opinion of the investigator, would pose an unacceptable risk to the subject; the subject is unable to meet the protocol requirement; will interfere with evaluation of investigational vaccine.
* Women who were breastfeeding or pregnant during the clinical study or planned to become pregnant during the study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-07-19 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse reactions (ARs) | Day 0-7 days after each vaccination
  The incidence of adverse reactions (ARs) within 7 days after each vaccination

SECONDARY OUTCOMES:
The occurrence of adverse events | Day 0-28 days after each vaccination
  The occurrence of adverse events within 28 days after vaccination
The incidences of serious adverse events (SAEs) and adverse events of special interest (AESIs) | Day 0 to 12 months after dose1, dose2 and dose 3.
  The incidences of serious adverse events (SAEs) and adverse events of special interest (AESIs) within 12 months after dose1, dose2 and dose 3.
Laboratory safety measures: coagulation, blood biochemistry, complete blood count and urinalysis | Day 3 after each vaccination.
  The change of laboratory safety measures on day 3 after each vaccination in comparison with that before vaccination.
Geometric neutralizing titers (GMT) of neutralizing antibody against SARS-CoV-2 wild strain and variants of concern(VOCs). | Day 14 after the second dose, day 14 , day 28 ,month 3, month 6, month 12 after full vaccination.
  GMT of neutralizing antibody against SARS-CoV-2 wild strain and variants of concern(VOCs) at day 14 after the second dose, day 14 ,day 28 , month 3, month 6, month 12 after full vaccination.
Geometric mean fold rise(GMFR) of neutralizing antibody against SARS-CoV-2 wild strain and variants of concern(VOCs). | Day 14 after the second dose, day 14, day 28, month 3, month 6, month 12 after full vaccination.
  GMFR of neutralizing antibody against SARS-CoV-2 wild strain and variants of concern(VOCs) at day 14 after the second dose, day 14 ,day 28, month 3, month 6, month 12 after full vaccination.
Seroconversion rate of neutralizing antibody against SARS-CoV-2 wild strain and variants of concern(VOCs). | Day 14 after the second dose, day 14, day 28, month 3, month 6, month 12 after full vaccination.
  Seroconversion rate of neutralizing antibody against SARS-CoV-2 wild strain and variants of concern(VOCs) at day 14 after the second dose, day 14 ,day 28, month 3, month 6, month 12 after full vaccination.
GMT of binding antibody against S protein of SARS-CoV-2 wild strain. | Day 14 after the second dose, day 14, day 28, month 3, month 6, month 12 after full vaccination.
  GMT of binding antibody against S protein of SARS-CoV-2 wild strain at day 14 after the second dose, day 14 ,day 28, month 3, month 6, month 12 after full vaccination.
GMFR of binding antibody against S protein of SARS-CoV-2 wild strain. | Day 14 after the second dose, day 14, day 28, month 3, month 6, month 12 after full vaccination.
  GMFR of binding antibody against S protein of SARS-CoV-2 wild strain at day 14 after the second dose, day 14 ,day 28, month 3, month 6, month 12 after full vaccination.
Seroconversion rate of of binding antibody against S protein of SARS-CoV-2 wild strain. | Day 14 after the second dose, day 14, day 28, month 3, month 6, month 12 after full vaccination.
  Seroconversion rate of binding antibody against S protein of SARS-CoV-2 wild strain at day 14 after the second dose, day 14 ,day 28, month 3, month 6, month 12 after full vaccination.
The cytokine levels (Elispot): Th1 type: IL-2, IFN-γ; Th2 type: IL-4. | Day 14 after the second dose, day 14 after full vaccination.
  The cytokine levels (Elispot) at day 14 after the second dose, day 14 after full vaccination.

OTHER OUTCOMES:
Anti-VLP antibody levels | Day 14, day 28, month 3, month 6, month 12 after full vaccination.
  Anti-VLP antibody levels at day 14, day 28, month 3, month 6, month 12 after full vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Fengcai Zhu, Principal Investigator — Jiangsu Provincial Center for Disease Control and Prevention
Locations (1):
- Jiangsu Provincial Center for Disease Control and Prevention, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tang R, Zeng Y, Zhou Y, Liang Q, Kang W, Yang Z, Zheng X, Zang X, Pan H, Jin J, Zhu F. Safety and immunogenicity of the SARS-CoV-2 LYB001 RBD-based VLP vaccine (CHO cell) phase 1 in Chinese adults: a randomized, double-blind, positive-parallel-controlled study. Expert Rev Vaccines. 2024 Jan-Dec;23(1):498-509. doi: 10.1080/14760584.2024.2337051. Epub 2024 May 2. PMID 38695310